CLINICAL TRIAL: NCT00210405
Title: Assessing the Feasibility and Effectiveness of Distributing Micronutrient Sprinkles Within a Title II Food Aid and Maternal and Child Health Program in Rural Haiti
Brief Title: Feasibility and Effectiveness of Distributing Micronutrient Sprinkles to Reduce Prevalence of Anemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Food Policy Research Institute (Other)
Collaborators: Cornell University (Other); World Vision (Other); Micronutrient Initiative (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-0460-INTFOO-01-3-IFPRI
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Anemia
Keywords: Anemia; Infant nutrition; Dietary supplements; Randomized controlled trials; Evaluation studies; Haiti
MeSH Terms: conditions — Anemia | interventions — Educational Status

ARMS (2):
- Food aid only (Active Comparator): Children in this arm received fortified food aid commodities supplied through the maternal and child health and nutrition program implemented by World Vision. They received fortified corn-soy blend, which contained iron.
  Interventions: Dietary Supplement: Fortified food aid (corn-soy blend)
- Micronutrient sprinkles + food aid (Experimental): Children in this arm were enrolled in the food assisted program, and therefore received fortified food aid, as well as 60 sachets of a multiple micronutrient powder (Sprinkles) containing iron, zinc, vitamin A, vitamin C and folic acid
  Interventions: Dietary Supplement: "Sprinkles" containing mulitple micronutrients; Behavioral: Education/communication on use of micronutrient sprinkles; Dietary Supplement: Fortified food aid (corn-soy blend)

INTERVENTIONS:
Dietary Supplement: "Sprinkles" containing mulitple micronutrients
  Arms: Micronutrient sprinkles + food aid
Behavioral: Education/communication on use of micronutrient sprinkles
  Arms: Micronutrient sprinkles + food aid
Dietary Supplement: Fortified food aid (corn-soy blend) — This intervention was part of the overall food assisted maternal and child health and nutrition program, and included fortified food aid commodities. Corn soy blend was targeted to the child, while the family also received wheat, lentils and oil.

SUMMARY:
The objective of this study is to test the feasibility and effectiveness of distributing micronutrient sprinkles to 6-20 month old children participating in an integrated maternal and child health and nutrition program in rural Haiti. The micronutrient sprinkles have been formulated to prevent or treat anemia in 6-23 month old children. Effectiveness in reducing the prevalence of anemia will be assessed.

DETAILED DESCRIPTION:
Anemia is highly prevalent among infants and young children in Haiti and throughout the world. Low intakes of several micronutrients contribute to this problem. It is very difficult to meet the micronutrient needs of infants and young children without substantial amounts of animal-source foods; such foods are not affordable for most families in many poor communities.

Micronutrient sprinkles are a novel approach to meeting children's needs. The sprinkles are packed in sachets containing a daily ration, and are intended to be used in the home and "sprinkled" directly on the children's food. Earlier trials have shown the efficacy of the sprinkles for preventing and treating anemia under controlled conditions.

The current study tests the feasibility and effectiveness when sprinkles are distributed in the programmatic context of a US Title II food aid distribution program, a context that is common in many countries that receive assistance from the United States Agency for International Development and other donors. The study also includes the development and dissemination of educational messages to motivate and enable caregivers to use the sprinkles properly. Based on previous efficacy trials no side-effects are anticipated, but the study also monitors for unanticipated side-effects.

Comparison: Since effectiveness of the sprinkles distributed as part of a take-home ration has not been established, this study employed a randomized controlled design. Randomization occurred at the level of the food distribution point (place where community members gather to receive food rations). Groups were assigned to receive either the take home ration (usual program practice) or the take home ration and the sprinkles. Families receiving only food rations at the control sites will receive sprinkles along with their food ration immediately after data collection is complete. The design was also consistent with the program necessity of a gradual roll-out of this new intervention. The prevalence of anemia among target-age children will be compared between groups that receive a two-month supply of micronutrient sprinkles with their take-home food ration, and those that do not.

ELIGIBILITY:
Inclusion Criteria:

* 6-20 months old at time of recruitment
* Family receives food rations at World Vision-Haiti's Food Distribution Points

Exclusion Criteria:

* Severe anemia at time of recruitment (hemoglobin <7.0 g/dl)

Ages: 6 Months to 20 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 450 (Actual)
Dates: Start 2005-03; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Prevalence of anemia after 2 months of treatment

SECONDARY OUTCOMES:
Prevalence of symptoms of morbidity at 1 and 2 months after treatment begins

CONTACTS AND LOCATIONS:
Overall Officials: Marie T. Ruel, PhD, Principal Investigator — International Food Policy Research Institute; Purnima Menon, PhD, Principal Investigator — International Food Policy Research Institute
Locations (1):
- World Vision-Haiti Regional Office, Hinche, Haiti

REFERENCES:
- [Background] Ruel MT, Menon P, Loechl C, Pelto G. Donated fortified cereal blends improve the nutrient density of traditional complementary foods in Haiti, but iron and zinc gaps remain for infants. Food Nutr Bull. 2004 Dec;25(4):361-76. doi: 10.1177/156482650402500406. PMID 15646314
- [Background] Zlotkin S, Arthur P, Schauer C, Antwi KY, Yeung G, Piekarz A. Home-fortification with iron and zinc sprinkles or iron sprinkles alone successfully treats anemia in infants and young children. J Nutr. 2003 Apr;133(4):1075-80. doi: 10.1093/jn/133.4.1075. PMID 12672922
- [Result] Menon P, Ruel MT, Loechl CU, Arimond M, Habicht JP, Pelto G, Michaud L. Micronutrient Sprinkles reduce anemia among 9- to 24-mo-old children when delivered through an integrated health and nutrition program in rural Haiti. J Nutr. 2007 Apr;137(4):1023-30. doi: 10.1093/jn/137.4.1023. PMID 17374671
- [Result] Loechl CU, Menon P, Arimond M, Ruel MT, Pelto G, Habicht JP, Michaud L. Using programme theory to assess the feasibility of delivering micronutrient Sprinkles through a food-assisted maternal and child health and nutrition programme in rural Haiti. Matern Child Nutr. 2009 Jan;5(1):33-48. doi: 10.1111/j.1740-8709.2008.00154.x. PMID 19161543
- See also: Sprinkles Global Health Initiative — http://sghi.org/about_sprinkles/index.html